CLINICAL TRIAL: NCT03641222
Title: A Non-Inferiority Randomized Controlled Trial Comparing Community (Group) Acupuncture to Individual Acupuncture to Alleviate Cancer Pain
Brief Title: Group Versus Individual Acupuncture for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Linda E. Carlson, Professor, Department of Oncology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-17-0237
Record Dates: First submitted 2018-07-10; First posted 2018-08-21 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Cancer; Pain
Keywords: Acupuncture; Group; Community Based; Individual; Randomized
MeSH Terms: conditions — Neoplasms; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Acupuncture (Experimental): Group acupuncture sessions take place in a multipurpose room, with 3-6 participants, each session lasts 30-45 minutes, occurring twice-weekly, over the course of six weeks, for a total of twelve treatments. The acupuncture was administered by a Naturopathic Doctor.
  Interventions: Device: Acupuncture
- Individual Acupuncture (Active Comparator): Individual acupuncture sessions take place in a multipurpose room, privately each session lasts 30-45 minutes, occurring twice-weekly, over the course of six weeks, for a total of twelve treatments. The acupuncture was administered by a Naturopathic Doctor.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Traditional Chinese Medicine (TCM) Acupuncture

SUMMARY:
Typically, in North America, acupuncture is performed on an individual basis. However, community acupuncture, also known as group acupuncture, is an emerging method of treating patients. Cancer patients, post-treatments were given acupuncture treatments to help alleviate pain, in a two-arm randomized trial.

DETAILED DESCRIPTION:
Typically, in North America, acupuncture is performed on an individual basis. However, community acupuncture, also known as group acupuncture, is an emerging method of treating patients. Although the practice can vary, community acupuncture is performed in a group setting, typically with reclining chairs dispersed around a large room, and one practitioner treating up to six people per session.

The outcomes of this this randomized controlled trial will allow the researchers to assess whether group acupuncture is a viable treatment option for people with cancer who are suffering from pain, especially those who are either resistant to or looking to avoid the side effects of opioids.

Objectives Examine the efficacy of community acupuncture for alleviating cancer pain, fatigue, sleep disturbances and distress when compared to individual acupuncture.

Evaluate the cost-effectiveness of community acupuncture compared to individual acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Adult cancer patients (≥18 years old), both male and female.
2. Experiencing pain with a minimum worst pain score (in the previous week) ≥3 on the 10-point Brief Pain Inventory (BPI).
3. All tumor groups, including metastatic patients.
4. Participant's pain can originate from any source, including postoperative, malignancy related, and neuropathic pain.
5. Must be willing to be randomized into either group, and must be able to attend a minimum of nine treatment sessions within a six-week period.

Exclusion Criteria:

1. Use of acupuncture within the previous six months.
2. Currently on or within one-month of active treatment (chemotherapy or radiation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The Brief Pain Inventory-Short Form | 6 weeks
  The Brief Pain Inventory-Short Form (BPISF) is a widely used self-report measure, originally developed for cancer pain, which measures both pain severity and pain interference

SECONDARY OUTCOMES:
The Profile of Mood States-Short Form | 6 weeks
  The Profile of Mood States-Short Form (POMS-SF) is a validated measure of psychological distress, which calculates Total Mood Disturbance (TMD) using six subscales: fatigue, vigor, tension, depression, anger and confusion (Shacham, 1983). The 37-item questionnaire asks patients to rate how various adjectives relate to how they have felt in the past week, on a Likert scale from zero (not at all) to four (extremely).
Pittsburg Sleep Quality Index | 6 weeks
  The Pittsburg Sleep Quality Index (PSQI) is 19-item questionnaire that measures quality of sleep and sleep disturbances
The Functional Assessment of Cancer Therapy-General | 6 weeks
  The Functional Assessment of Cancer Therapy-General (FACT-G) is a 20-item questionnaire that measures health-related quality of life (HRQOL) within the cancer population. The questionnaire contains four subscales: physical, social/family, emotional and functional well-being.
The Functional Assessment of Cancer Therapy - Fatigue | 6 weeks
  The Functional Assessment of Cancer Therapy-Fatigue (FACT-F) comprised of the FACT-G, plus an additional 13 questions related to fatigue
The Inventory of Socially Supportive Behaviours | 6 weeks
  The Inventory of Socially Supportive Behaviours (ISSB) Short Form is an 18-item questionnaire designed to measure social support, which asks participants to indicate the number of times they have experienced particular behaviours in the past month
Edmonton Symptom Assessment Scale | 6 weeks
  The Edmonton Symptom Assessment Scale (ESAS) is a simple screening measure that can be used to assess various physical and psychological symptoms, originally designed for palliative care patients
A Pain Visual Analog Scale | 6 weeks
  The pain visual analog scale (VAS) consists of a 10 centimetre line on a slip of white paper, with the indicators "no pain at all" on the far-left end, and "worst pain imaginable" on the far-right end
The European Quality of Life-5 Dimensions | 6 weeks
  This utility scoring instrument is intended to provide an overall quality of life evaluation with a scale from 1 (perfect health) to 0 (death) and allows for the calculation of quality adjusted life years (QALYs)

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Carlson, PhD, Principal Investigator — University of Calgary
Locations (1):
- Psychosocial Oncology, Cancer Control Alberta, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oberoi D, Reed EN, Piedalue KA, Landmann J, Carlson LE. Exploring patient experiences and acceptability of group vs. individual acupuncture for Cancer-related pain: a qualitative study. BMC Complement Med Ther. 2022 Jun 13;22(1):155. doi: 10.1186/s12906-022-03600-6. PMID 35698124
- [Derived] Oberoi DV, Longo CJ, Reed EN, Landmann J, Piedalue KL, Carlson LE. Cost-Utility of Group Versus Individual Acupuncture for Cancer-Related Pain Using Quality-Adjusted Life Years in a Noninferiority Trial. J Altern Complement Med. 2021 May;27(5):390-397. doi: 10.1089/acm.2020.0386. Epub 2021 Apr 27. PMID 33904784
- [Derived] Oberoi D, McLennan A, Piedalue KA, Wayne PM, Jones JM, Carlson LE. Factors Influencing Preference for Intervention in a Comparative Effectiveness Trial of Mindfulness-Based Cancer Recovery and Tai Chi/Qigong in Cancer Survivors. J Altern Complement Med. 2021 May;27(5):423-433. doi: 10.1089/acm.2020.0400. Epub 2021 Apr 27. PMID 33902334